CLINICAL TRIAL: NCT04356547
Title: Orotracheal Intubation Using Flexible Fibro Bronchoscope With vs Without Supraglottic Device AuraGain in Pediatric Simulators: Cross Over Clinical Trial
Brief Title: Orotracheal Intubation Using Flexible Fibro Bronchoscope With vs Without Supraglottic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Mario Zamudio, Clinical Professor, Universidad de Antioquia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: F-017-00
Record Dates: First submitted 2020-02-05; First posted 2020-04-22 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Intubation;Difficult
Keywords: Fiberoptic intubation; Pediatrics; laryngeal mask; Intubation, intratracheal; Manikins
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Intervention Model Description: The study will be a controlled, cross-sectional, randomized, non-blind, superiority trial and will be realized in a simulation center, with pediatric manikins. It includes 41 anesthesiologists or anesthesiology residents, who will be randomized to start their participation in the clinical trial in the intervention or control group. Subsequently, they will become part of the opposing group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiberoptic intubation using laryngeal mask AuraGain (Active Comparator): Participants should perform an fiberoptic tracheal intubation through the AuraGain laryngeal mask, in a pediatric simulator. Will be evaluated the success rate at the first attempt and other secondary outcomes
  Interventions: Device: Fiberoptic intubation with laryngeal mask AuraGain
- Fiberoptic intubation without laryngeal mask (Active Comparator): Participants should perform an fiberoptic tracheal intubation without laryngeal mask, in a pediatric simulator. Will be evaluated the success rate at the first attempt and other secondary outcomes
  Interventions: Device: Fiberoptic intubation without laryngeal mask

INTERVENTIONS:
Device: Fiberoptic intubation with laryngeal mask AuraGain — Participants should perform an fiberoptic tracheal intubation through the AuraGain laryngeal mask, in a pediatric simulator.
  Arms: Fiberoptic intubation using laryngeal mask AuraGain
Device: Fiberoptic intubation without laryngeal mask — Participants should perform an fiberoptic tracheal intubation without laryngeal mask, in a pediatric simulator.
  Arms: Fiberoptic intubation without laryngeal mask

SUMMARY:
Randomized clinical trial conducted in pediatric simulators that wishes to compare the success of fiberoptic tracheal intubation using supraglottic device AuraGain compared with fiberoptic tracheal intubation without laryngeal mask, performed by anesthesiologists and anesthesiology residents.

DETAILED DESCRIPTION:
To determine the required sample size, the data reported from studies were studied where the Auragain device for intubation with fibrobronchoscope in adult patients is studied. In these studies, an average intubation rate at the first attempt in adults of 87% of all cases was found compared to an average success rate of intubation with FBC without a supraglottic device of 60%. Based on these data, and assuming an alpha error of 0.05 of two tails and a power of 80%, a total number of participants of 82 is required, that is 41 participants per group. However, being a cross study, a total of 41 participants is required since each participant will be their own control. For its calculation, the Stata 14.0 program was used Sample size

Recruitment The recruitment of participants will be carried out by the research group. A verbal and email invitation will be made to the anesthesiology residents from different University centers, in addition to the residents of this same specialty of other institutions that are doing some rotation at the University Hospital San Vicente Foundation or IPS University Clinic León XIII. In the same way the anesthesiologists of these two health institutions will be recruited for the study.

Sampling will be carried out for the convenience of consecutive participants until the necessary number is fulfilled according to the sample design.

After this, the possible participants of the clinical trial will be asked about their intention to be part of the study, and those interested will be explained the relevant aspects of this study, including the protocol, objectives, safety aspects and doubts will be resolved.

Once they accept their participation in the clinical trial, the eligibility criteria to enter the study will be determined and it will be remembered that they must perform a CUSUM learning curve for fibrobronchoscopy in pediatric simulators. If the participant accepts the informed consent, authorizing the proceeding of the study.

A recruitment rate of 4 to 5 participants per week is expected, so a recruitment period of 10 weeks after study approval is calculated.

The strategies used to favor recruitment will be:

* Create a work team with interest in the area and committed to the development of the study.
* Motivate residents of anesthesiology and anesthesiologists through information boards in the operating rooms of the San Vicente Foundation University Hospital or IPS University Clinic León XIII
* Perform a check every two weeks to determine that recruitment goals are being met

It should be clarified that there will be no economic incentive for the patients or the group of anesthesiologists participating in the study Retention The participants understudy do not participate in economic stimulation that the incentives to participate or continue in. Participation will be voluntary, free acceptance of the anesthesiologist or anesthesiology student, who has understood the scientific benefits of the study and the possible associated risks.

Losses: Participants who perform the intervention or control and the selected data will be evaluated immediately after intubation maneuvers. There will be no subsequent measurements that involve the monitoring of the participants. It is unlikely that participants will be lost since data collection is immediate, however, and given that complications occur at different times, there is a the possibility that the participant does not attend one or both moments of intervention so a loss of 5% of participants is projected.

Withdrawals: Since all participants will be trained with the CUSUM curve, there are no causes to withdraw participants, the only cause will be that the participant will not wish to continue the investigation once the informed consent has been completed. In case this happens by sending a written report to the research coordinator.

Analysis by intention to be treated: Due to the nature of the study, participants can perform intubation maneuvers with both arms, see this type of analysis by default.

Data management

The plan for handling data, inputs, coding, security, and storage, which guarantee their quality will be as follows:

* Collection: The researcher who observes the intervention of the participant will record the data in physical format, then the data recorded in the physical formats will be subjected to quality control; avoiding loss and error in data entry. This information will be subject to review by double-checking by two different investigators.
* Sending of the data: Once the data has been collected, they are entered into an envelope, marked according to the assignment number and the participant's identification number, and sealed. They will be sent to the data collection center, located in the Anesthesiology and Resuscitation Section office.
* Coding: The data will be entered in a magnetic medium (Excel © 2010) by an assistant of the research group, who does not participate in the research directly. A second assistant performs the double-check, to verify the agreement between the data entered and the data reported.
* Security: It will be encrypted with a password that only the auxiliaries who collect the data know. Periodically, the assistants will take a backup to keep the data, with restricted access for researchers.
* Storage: Envelopes with the information of physical formats will be stored for 2 years after the end of the study in the office of Anesthesiology and Resuscitation Section.
* Analysis: Once the collection stage is finished and the analysis begins, the data will be delivered to the researchers with allocation concealment.

  18. Statistical method and Analysis Plan. The baseline characteristics will be presented in Table 1. For quantitative variables, Shapiro Wills normality test will be performed, and if they are normal, they will be presented by means and standard deviation; if normality is not demonstrated, they will be presented through medians and interquartile range. For qualitative variables, it will be presented by frequencies and proportions.

The results will be presented at relative risk with their respective 95% confidence interval, with the value of p, so Fisher's exact test will be performed. A p-value of less than 0.05 will be considered statistically significant.

For the other outcomes, the statistical analysis will be presented (Outcome, Measures, and methods of analysis):

Intubation success at first attempt: Incidents Relative Risk Fisher's exact test.

Time in seconds of the intubation maneuver : Mean or median, Difference of means or medians Student t-test or Mann Whitney U test. In case of non-normality in this variable, it will be considered to report in the median and a non-parametric test will be carried out as a hypothesis test.

Global intubation successful: Incidents, Relative Risk Fisher's exact test

Display Degree: Proportion of each grade Relative Risk Chi-square test of homogeneity

Intubation success at the second and third attempt: Incidents Relative Risk Fisher's exact test

Accidental extubation: Incidents Relative Risk Fisher's exact test Degree of the difficulty of orotracheal intubation: Proportion of each grade Relative Risk Chi-square test of homogeneity

Analysis of lost data

Due to the nature of the study, participants will perform intubation maneuvers in both arms, so it is not possible to perform this type of analysis. A loss should not occur, as the data will be collected immediately, except in cases of force majeure. Methods of the imputation of lost data will not be used.

Data monitoring and interim analysis.

The data monitoring will be carried out by the external research committee consisting of 2 anesthesiologists from the Department of Anesthesiology and Resuscitation of the University of Antioquia and staff of the research institute of the same higher education institutions. They will have as function:

1. Evaluation and monitoring of recruitment, randomization, adherence to the protocol, among others.
2. Blindly evaluate and monitor research data and generate recommendations to the research group. Among the suggested recommendations may be the suspension of the investigation.
3. Interim analysis: They will not be carried out, because the study will be carried out in simulators, no serious adverse effects are planned and the recruitment time is not prolonged.

Audit

The data quality audit will be carried out by a person from the Anaesthesiology and Resuscitation service, who will have the function of:

1. Evaluate the the relevance of data collection formats and databases designated for the registration of information.
2. Evaluate adherence to the protocol by researchers.
3. An audit will be conducted after the end of the third week of recruitment, taking as a sample the data of 50% of participants who have entered the study.

The research team must adopt the following measures to guarantee the quality of data management:

1. Develop a procedure manual that is easily accessible to researchers, with availability in the simulation service, which clearly states the objectives, eligibility criteria, outcomes, randomization, and diligence of informed consent.
2. Data collection formats: that contain clear information and that are agile to complete.
3. Training and evaluation of the research team to ensure homogeneity in the application of the protocol.
4. Double review of the data that is transferred from the physical medium to the magnetic medium. Storage of physical data to be reviewed in case of loss of data in electromagnetic media.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists or anesthesiology residents
* Perform a training in fiber optic tracheal intubation whit and without supraglottic device in simulators. The CUSUM learning curve will be used to achieve a success rate greater than 80% at the first attempt.
* Accept to participate in the study and sign the informed consent

Exclusion Criteria:

* Not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Successful intubation at the first attempt using fiber optic through laryngeal mask AuraGain compared to fiberoptic intubation without laryngeal mask | immediately after intubation
  Incidence of successful tracheal intubation at the first attempt using fiberoptic through laryngeal mask AuraGain and without laryngeal mask. After this procedure, tracheal intubation with positive pressure ventilation in the pediatric simulators will be verified.

SECONDARY OUTCOMES:
Time required to achieve tracheal intubation using fiber optic through laryngeal mask AuraGain compared to fiberoptic intubation without laryngeal mask | immediately after intubation
  The seconds needed from the moment the participant takes the fibroscope with their hands until the first ventilation is achieved with positive pressure.
Successful intubation at the second and third attempts using fiber optic through laryngeal mask AuraGain compared to fiberoptic intubation without laryngeal mask | immediately after intubation
  Incidence of successful tracheal intubation at the second and third attempts using fiberoptic through laryngeal mask AuraGain and without laryngeal mask. After this procedure, tracheal intubation with positive pressure ventilation in the pediatric simulators will be verified
Global success of orotracheal intubation using fiber optic through laryngeal mask AuraGain compared to fiberoptic intubation without laryngeal mask | immediately after intubation
  Global success is considered when tracheal intubation is achieved regardless of the number of attempts. The maximum number of attempts in each group is 3.
Accidental extubation at the time of removing the bronchoscope and/or the laryngeal mask. | immediately after intubation
  Incidence of accidental extubation at the time of removing the laryngeal mask or fiber optic bronchoscope will be evaluated by the lack of ventilation with positive pressure after achieving successful tracheal intubation in pediatric simulators
Ease of tracheal intubation | immediately after intubation
  The subjective scale of ease to achieve tracheal intubation. It is a scale from 0 to 10, where 0: extremely difficult and 10: extremely easy.
Degree of glottic visualization | immediately after intubation
  Glottic display scale. Class 1: Unable to see the vocal cords. Class 2: the vocal cords and the anterior aspect of the epiglottis are visualized. Class 3: the vocal cords and the posterior aspect of the epiglottis are observed. Grade 4: only vocal cords were observed.

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Zamudio, Professor, Principal Investigator — Universidad de Antioquia
Locations (2):
- Colombia (2):
  - Mario Andres Zamudio, Medellín, Antioquia
  - Antioquia´s University, Medellín

IPD SHARING:
Plan to Share IPD: Yes
The data will be stored for future research in the database of the GRIMPA perioperative medicine research group
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5 years
Access Criteria: Formal application and authorization of the University of Antioquia